CLINICAL TRIAL: NCT00026156
Title: Phase II Trial of Sequential Vinorelbine and Docetaxel in Advanced Non-Small Cell Lung Cancer Patients Age Seventy and Older, or With Performance Status 2
Brief Title: S0027: Vinorelbine Followed by Docetaxel in Treating Patients With Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068991; S0027 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2001-11-09; First posted 2003-01-27 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; squamous cell lung cancer; large cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; adenocarcinoma of the lung
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung | interventions — Docetaxel; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: docetaxel
Drug: vinorelbine tartrate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of vinorelbine followed by docetaxel in treating patients who have advanced non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the survival of patients with advanced non-small cell lung cancer who are either age 70 and over or who have performance status 2, when treated with sequential vinorelbine and docetaxel. (Age 70 and older with Zubrod 0-1 stratum closed to accrual as of 2/15/2003.)
* Determine the objective tumor response rates, including confirmed and unconfirmed and complete and partial, in patients treated with this regimen.
* Assess the dose delivered and the reported functional symptom status of patients treated with this regimen.
* Determine the toxic effects of this regimen in these patients.
* Determine the feasibility of performing pharmacokinetic studies and obtaining pharmacokinetic data on these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to age and performance status (age 70 and over with Zubrod 0-1 vs age 18 and over with Zubrod 2). (Age 70 and older with Zubrod 0-1 stratum closed to accrual as of 2/15/2003.)

Patients receive vinorelbine IV over 6-10 minutes on days 1 and 8. Treatment repeats every 21 days for 3 courses in the absence of unacceptable toxicity. Beginning 2 weeks after the last dose of vinorelbine, patients receive docetaxel IV over 1 hour on days 1, 8, and 15. Treatment repeats every 28 days for 3 courses in the absence of unacceptable toxicity.

Quality of life is assessed at baseline, at the beginning of courses 2-6, and at week 22.

Patients are followed at week 22, every 3 months for 1 year, and then every 6 months for 2 years.

PROJECTED ACCRUAL: A minimum of 95 patients (55 patients age 70 and over with Zubrod 0-1 and 40 patients age 18 and over with Zubrod 2) will be accrued for this study within 12-18 months. (Age 70 and older with Zubrod 0-1 stratum closed to accrual as of 2/15/2003.)

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed, newly diagnosed, advanced primary non-small cell lung cancer (NSCLC) (adenocarcinoma, large cell carcinoma, squamous cell carcinoma, or unspecified), designated as 1 of the following stages:

  * Selected stage IIIB (excluding Pancoast tumors)

    * T4 lesion due to malignant pleural effusion OR
    * Multiple lesions in a single lobe containing a T3 or T4 primary
  * Stage IV (any T, any N, M1)
  * Recurrent disease after prior surgery and/or radiotherapy
* Measurable or evaluable disease outside of prior radiation port
* No bronchoalveolar carcinoma
* No brain metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Zubrod 0-1 (for age 70 and over) (Age 70 and older with Zubrod 0-1 stratum closed to accrual as of 2/15/2003)
* Zubrod 2 (for age 18 and over)

Life expectancy:

* Not specified

Hematopoietic:

* Absolute granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than upper limit of normal (ULN)
* SGOT/SGPT no greater than 2 times ULN if alkaline phosphatase is no greater than ULN OR
* Alkaline phosphatase no greater than 4 times ULN if SGOT/SGPT are no greater than ULN

Renal:

* Not specified

Other:

* No prior severe hypersensitivity to docetaxel or other drugs formulated with polysorbate 80
* No grade 2 or greater sensory neuropathy
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or other adequately treated stage I or II cancer in complete remission
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior or concurrent biologic therapy for NSCLC
* No concurrent filgrastim (G-CSF)

Chemotherapy:

* No prior systemic chemotherapy for NSCLC

Endocrine therapy:

* No prior or concurrent hormonal therapy for NSCLC

Radiotherapy:

* See Disease Characteristics
* At least 3 weeks since prior radiotherapy and recovered
* Concurrent palliative radiotherapy to small-field nonmeasurable lesions (i.e., painful bony lesions) allowed
* No other concurrent radiotherapy

Surgery:

* See Disease Characteristics
* At least 3 weeks since prior thoracic or other major surgery and recovered

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2001-11; Primary Completion 2004-07 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul J. Hesketh, MD, Study Chair — Steward St. Elizabeth's Medical Center of Boston, Inc.
Locations (96):
- United States (96):
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - Veterans Affairs Medical Center - Phoenix (Carl T. Hayden), Phoenix, Arizona
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Veterans Affairs Medical Center - Little Rock (McClellan), Little Rock, Arkansas
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Veterans Affairs Medical Center - West Los Angeles, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Veterans Affairs Outpatient Clinic - Martinez, Martinez, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Davis Cancer Center, Sacramento, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - David Grant Medical Center, Travis Air Force Base, California
  - University of Colorado Cancer Center, Denver, Colorado
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - MBCCOP - Howard University Cancer Center, Washington D.C., District of Columbia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Dwight David Eisenhower Army Medical Center, Fort Gordon, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - MBCCOP - University of Illinois at Chicago, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - Veterans Affairs Medical Center - Hines (Hines Junior VA Hospital), Hines, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Genesis Medical Center, Davenport, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - MBCCOP - LSU Medical Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - St. Elizabeth's Medical Center, Boston, Massachusetts
  - Veterans Affairs Medical Center - Boston (Jamaica Plain), Jamaica Plain, Massachusetts
  - Veterans Affairs Medical Center - Ann Arbor, Ann Arbor, Michigan
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - CCOP - Beaumont, Royal Oak, Michigan
  - Providence Hospital - Southfield, Southfield, Michigan
  - Veterans Affairs Medical Center - Biloxi, Biloxi, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Veterans Affairs Medical Center - Jackson, Jackson, Mississippi
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Veterans Affairs Medical Center - Albuquerque, Albuquerque, New Mexico
  - MBCCOP - University of New Mexico HSC, Albuquerque, New Mexico
  - Veterans Affairs Medical Center - Albany, Albany, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Veterans Affairs Medical Center - Cincinnati, Cincinnati, Ohio
  - Barrett Cancer Center, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Veterans Affairs Medical Center - Oklahoma City, Oklahoma City, Oklahoma
  - Veterans Affairs Medical Center - Portland, Portland, Oregon
  - CCOP - Columbia River Program, Portland, Oregon
  - Oregon Cancer Institute, Portland, Oregon
  - Veterans Affairs Medical Center - Charleston, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - University of Tennessee Cancer Institute, Memphis, Tennessee
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Veterans Affairs Medical Center - Houston, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - Veterans Affairs Medical Center - Temple, Temple, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Veterans Affairs Medical Center - Salt Lake City, Salt Lake City, Utah
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington

REFERENCES:
- [Background] Hesketh PJ, Lilenbaum RC, Chansky K, Dowlati A, Graham P, Chapman RA, Crowley JJ, Gandara DR. Chemotherapy in patients > or = 80 with advanced non-small cell lung cancer: combined results from SWOG 0027 and LUN 6. J Thorac Oncol. 2007 Jun;2(6):494-8. doi: 10.1097/JTO.0b013e318060097e. PMID 17545843
- [Result] Hesketh PJ, Chansky K, Lau DH, Doroshow JH, Moinpour CM, Chapman RA, Goodwin JW, Gross HM, Crowley JJ, Gandara DR. Sequential vinorelbine and docetaxel in advanced non-small cell lung cancer patients age 70 and older and/or with a performance status of 2: a phase II trial of the Southwest Oncology Group (S0027). J Thorac Oncol. 2006 Jul;1(6):537-44. PMID 17409914
- [Result] Hesketh PJ, Chansky K, Lau DH, et al.: Sequential vinorelbine (V) and docetaxel (D) in advanced non-small cell lung cancer (NSCLC) patients age > 70, or with performance status (PS) 2: a SWOG phase II trial (S0027). [Abstract] J Clin Oncol 22 (Suppl 14): A-7056, 630s, 2004.